CLINICAL TRIAL: NCT04909528
Title: Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Premature Ventricular Contractions
Brief Title: LLTS to Treat Premature Ventricular Contractions
Acronym: TREAT-PVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: University of Oklahoma (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Wuxi No. 2 People's Hospital (Other); The First People's Hospital of Changzhou (Other); Second Affiliated Hospital of Nantong University (Other); Affiliated Hospital of Nantong University (Other); Geriatric Hospital of Nanjing Medical University (Other); First Affiliated Hospital of Wannan Medical College (Other); Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-SR-328
Record Dates: First submitted 2021-05-19; First posted 2021-06-01 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Premature Ventricular Contraction
Keywords: Premature Ventricular Contraction; Low-level Tragus Stimulation; autonomic nerve modulation
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Low-level tragus stimulation
  Interventions: Device: Low-level tragus stimulation
- Control Group (Sham Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Low-level tragus stimulation — Frequency: 20Hz; Pulse width: 0.2 ms; Current is based on the following: Determine the perception threshold (feeling tingling) at the time of baseline information assessment. Because of sensory adaptation, ask the patient 5 minutes later to increase the current by 1-5 mA. Try to find the current level below the discomfort level and above the perception threshold; Stimulation spot: ear tragus; Stimulation time: 30 min in the morning (from 6:00 a.m. to 9:00 a.m.) and 30 min in the evening (from 20:00 p.m. to 23:00 p.m.)
  Arms: Experimental Group
Device: Sham stimulation — Frequency: 20 Hz; Pulse width: 0.2 ms; Current is based on the following: Determine the perception threshold (feeling tingling) at the time of baseline information assessment. Because of sensory adaptation, ask the patient 5 minutes later to increase the current by 1-5 mA. Try to find the current level below the discomfort level and above the perception threshold; Stimulate spot: ear lobe. Stimulation time: 30 min in the morning (from 6:00 a.m. to 9:00 a.m.) and 30 min in the evening (from 20:00 p.m. to 23:00 p.m.)
  Arms: Control Group

SUMMARY:
This randomized control trial is designed to explore the effect of low-level tragus stimulation in patients with frequent premature ventricular contractions.

DETAILED DESCRIPTION:
Background Premature ventricular contraction (PVC), also known as premature ventricular beat, is one of the most common symptomatic arrhythmias in clinical practice. PVCs may cause serious harm to patients as follow: 1. PVCs with considerable load can increase the incidence of cardiomyopathy; 2. Some recurrent malignant arrhythmias, such as ventricular tachycardia and ventricular fibrillation, can be induced by PVCs; 3. cardiac resynchronization therapy-pacing/defibrillator non-responders may be due to frequent PVCs, which reduce the proportion of biventricular pacing; 4. For structural heart disease patients, PVCs may make their damaged heart function further deteriorated. At present, the clinical treatment of PVCs is still based on drugs, such as beta-blockers, mexiletine, propafenone, etc., and their effectiveness varies greatly among individuals. The status of catheter ablation in the treatment of ventricular premature beats continuous improvement, but this is an invasive operation and relatively expensive, which limits its wide application in clinical practice. Recent studies have shown that the autonomic nervous system plays an important role in the occurrence and maintenance of ventricular arrhythmia. Relevant studies have confirmed that the onset of ventricular arrhythmia is related to sympathetic nerve excitement. Moreover, inhibiting sympathetic nerve activity, including anesthesia, sympathetic nerve block, sympathetic nerve denervation, etc., can effectively reduce the onset and burden of ventricular arrhythmia. On the other hand, in patients with myocardial ischemia-related ventricular arrhythmia, atrial arrhythmia, and heart failure, the safety and effectiveness of the treatment of vagus nerve stimulation have also been verified. Low-level tragus stimulation (LLTS) is an emerging method of regulating autonomic nerves. Functional cardiac magnetic resonance studies have confirmed that by stimulating the auricle branch of the vagus nerve distributed in the tragus of the outer ear, the central projection of the vagus nerve in the brainstem and other higher centers can be activated. It is worth noting that LLTS has been used in clinical practice to treat tinnitus and epilepsy. Moreover, recent studies have confirmed that LLTS can reduce sympathetic nerve activity, inhibit inflammatory factors, and reduce the atrial fibrillation burden in patients with paroxysmal atrial fibrillation.

Aim of the Study The current trial is designed to explore the effect of low-level tragus stimulation in patients with frequent premature ventricular contractions.

Study Design This is a randomized, prospective, parallel, single-blind multicenter design. The enrollment target for this investigation is 100 patients. Patients are randomized in a 1:1 fashion into one of the investigation arms: active and sham LLTS group. Active LLTSs are performed using a transcutaneous vagus nerve stimulation device (Parasym device, Parasym Health, London, United Kingdom) with an ear clip attached to the tragus of the right ear. In the sham group, the clips are attached to the ear lobe and regarded as effectless to vagus nerve. At baseline, 3 months, and 6 months, patients underwent noninvasive continuous ECG monitoring for 10 days to evaluate their PVC burden (deﬁned as the percentage of premature ventricular beats in total heart beats) using an adhesive continuous ECG patch. Heart rate variability, quality of life, skin sympathetic nerve activity and serum cytokine measurement are evaluated at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >18, <80 of age
* Symptomatic PVCs refractory to ≥1 antiarrhythmic drugs (including β-blockers and calcium-channel blockers).
* PVC burden ≥ 10%, with or without prior ablation
* Arrhythmias originated from any focus (foci) in the right ventricular or left ventricular.

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 45% unless proven to be PVC-mediated cardiomyopathy (history of improving LVEF by >15% when PVC burden was reduced by pharmacological agents or ablation)
* EF continues to decrease in the past 4 months regardless of the etiology
* Unwilling to continue current pharmacological therapy during the study period
* Severe heart failure with New York Heart Association Class ≥ III
* Ventricular arrhythmias attributed to underlying structural heart disease, known myocardial scar or myocarditis
* Change of anti-arrhythmic drug dosing, including β-blockers and calcium channel blockers, within 2 months prior to enrollment
* < 3 months after prior unsuccessful ablation:
* Patients on amiodarone
* Patients with known thyroid issues, on renal-dialysis
* life expectancy of < 12 months
* Sustained ventricular tachycardia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PVC burden | 3 months follow-up
  Patients underwent noninvasive continuous ECG monitoring using an adhesive continuous ECG patch for 10 days to evaluate their PVC burden which is deﬁned as the percentage of premature ventricular beats in total heart beats.
PVC burden | 6 months follow-up
  Patients underwent noninvasive continuous ECG monitoring using an adhesive continuous ECG patch for 10 days to evaluate their PVC burden which is deﬁned as the percentage of premature ventricular beats in total heart beats.

SECONDARY OUTCOMES:
Questionnaire to score severity of symptoms and quality of life | 3 months and 6 months follow-up
  Patients are required to complete 36-item short form health survey questionnaire to score severity of symptoms and quality of life. The scores ranges from 0-100. Higher scores mean healthier status.
Serum cytokine marker | 3 months and 6 months follow-up
  hsCRP (mg/L) level in serum
Serum cytokine marker | 3 months and 6 months follow-up
  Interleukin-6 (ng/mL) level in serum
Skin sympathetic nerve activity | 3 months and 6 months follow-up
  20-min recording using our customized device. The electrical activity that can be measured on the surface of the skin originates from the heart, the muscle or nerve structures. Because the frequency content of nerve activity falls in a higher frequency range than that of the ECG and myopotential, it is possible to use high-pass or band-pass ﬁltering to speciﬁcally isolate the skin sympathetic nerve activity. The unit of measure is µV.
Treatment compliance | 3 months and 6 months follow-up
  acquire patients' stimulation diaries to assess compliance
Number of participants with adverse effects | 3 months and 6 months follow-up
  Number of participants with pruritus, flush, pain at the stimulation cite
Heart rate variability | 3 months and 6 months follow-up
  Parameters include Standard deviation of the NN (R-R) intervals, Low frequency/High frequency ratio et al. which reflect sympathovagal balance and are calculated according to holter recording

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Cai C, Wu N, Yang G, Yang S, Liu W, Chen M, Po SS; TREAT PVC investigators. Transcutaneous electrical vagus nerve stimulation to suppress premature ventricular complexes (TREAT PVC): study protocol for a multi-center, double-blind, randomized controlled trial. Trials. 2023 Oct 23;24(1):683. doi: 10.1186/s13063-023-07713-2. PMID 37872628